CLINICAL TRIAL: NCT04360668
Title: Determining the Effect of a Combination of Muscle Energy Techniques and Trigger Point Therapy on Subjective and Objective Indicators Assessing the Condition of the Musculoskeletal System in Asymptomatic Persons With Latent Trigger Point
Brief Title: Muscle Energy Techniques and Trigger Point Therapy in Asymptomatic Persons With Latent Trigger Point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Michał Wendt, PhD, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PoznanUPhyEd
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Asymptomatic Condition
Keywords: muscle energy techniques; trigger point therapy; range of motion; soft tissue properties; pressure pain threshold; combination of therapeutic methods
MeSH Terms: conditions — Asymptomatic Diseases

STUDY DESIGN:
Intervention Model Description: The first stage will involve recruitment. 60 people will be gathered based on the qualifying and disqualifying criteria. This group of participants will be randomized. Each participant will draw a number that will determine the assignment to a specific group (MET plus TPT group, single MET or single TPT group). Preliminary measurements will be collected before the intervention. Each participant will have a specific intervention depending on which research group they belong to. The therapist will be responsible for performing the given therapeutic technique. Immediately after the intervention and on the second day, data will be collected by the researcher. The person conducting the function of coordinator will supervise the proper conduct of the scientific research. The collected data will be analyzed by the outcomes assessor.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not know which research group they will belong to. Each participant will draw a number that will be specific to the given research group. The investigator will also not know which group the participant belongs to (he will only use the participant's number). The outcomes assessor will not know which group is experimental and which are active comparators (they will be marked numerically instead of using a name). The correct course of the study will be supervised by a person who acts as a coordinator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Muscle Energy Technique combined with Trigger Point Therapy (Experimental): For this group of participants, combined therapy (Muscle Energy Technique with Trigger Point Therapy) will be used
  Interventions: Other: Muscle Energy Technique (MET) combined with Trigger Point Therapy (TPT)
- Muscle Energy Technique (Active Comparator): For this group of participants, a single method (Muscle Energy Technique) will be used
  Interventions: Other: Muscle Energy Technique (MET)
- Trigger Point Therapy (Active Comparator): For this group of participants, a single method (Trigger Point Therapy) will be used
  Interventions: Other: Trigger Point Therapy (TPT)

INTERVENTIONS:
Other: Muscle Energy Technique (MET) — The Contract-Relax Agonist-Contract (CRAC) technique will be used, which belongs to the broad MET group. The participant will be in the supine position. The therapist will set the cervical segment in the lateral flexion until a slight soft tissue tension is felt. The technique will consist of two stages. In the first phase (contraction phase), the upper trapezius will be activated against the therapist's resistance (shoulder girdle elevation) - 10 seconds. Then the person undergoing the procedure breathes in and out deeply. Then 10 seconds of antagonist group contraction (shoulder girdle depression) will be performed. Next, the therapist will passively move the participant's shoulder girdle towards the depression. Then the second phase will follow (stretching phase), during which the participant will passively lie in the back position for 30 seconds. Both phases will make up the therapeutic cycle. Each participant will have 5 cycles on each side of the upper trapezius.
  Arms: Muscle Energy Technique
Other: Trigger Point Therapy (TPT) — The technique of Positional Release (PR) will be used, which is one of the broadly understood Trigger Point Therapy. It will consist in compressing the trigger point with a simultaneous shortening of muscle attachments (slight lateral flexion towards the relaxed muscle). The muscle on both sides will be treated. The pressure exerted by the therapist's pincer grip will be acceptable to the patient. The duration of the technique will be 2 minutes for each muscle. While performing this technique, the participant will passively lie on his back.
  Arms: Trigger Point Therapy
Other: Muscle Energy Technique (MET) combined with Trigger Point Therapy (TPT) — For this type of intervention, TPT will first be performed on both sides of the upper trapezius muscle, followed by MET, which will also be performed bilaterally. The detailed method of performing the applied therapeutic techniques for the combined procedure will be identical as in the case of isolated (single) methods.
  Arms: Muscle Energy Technique combined with Trigger Point Therapy

SUMMARY:
The main objective of this study is to evaluate the effectiveness of therapy which will be a combination of Muscle Energy Technique (MET) and Trigger Point Therapy (TPT), performed bilaterally on the upper trapezius muscle in the group of asymptomatic persons with latent trigger point. The study will show whether one-time therapy has an impact on: mobility of the cervical spine, biophysical parameters (muscle tone, stiffness and elasticity) of soft tissues and pressure pain threshold of upper trapezius muscle. An additional goal will be to compare the effectiveness of the three treatments used: combination of MET with TPT, single MET and single TPT.

Research hypotheses:

* The combination of MET with TPT will increase the angular ranges of basic cervical spine movements immediately after the therapy and these effects will persist the second day after the intervention.
* The combination of MET with TPT will increase the elasticity and reduce muscle tone and stiffness in the area of the upper trapezius immediately after the therapy, and these effects will persist the second day after the intervention.
* The combination of MET with TPT will increase the pressure pain threshold of upper trapezius muscle immediately after the therapy, and this effect will persist the second day after the intervention.
* The combination of MET with TPT will be more effective than single MET and single TPT methods.

Muscle Energy Techniques (MET) can be defined as a group of soft tissue manipulation methods. They are a multi-task techniques that can be performed to improve the function of the musculoskeletal system and reduce pain. METs are used by clinicians who treat various myofascial and joint dysfunctions as well as a form of prevention and protection of the musculoskeletal system.

Trigger point therapy (TPT) uses manual techniques such as ischemic compression (IC), positional release (PR), dry needling and soft tissue manipulations [TP1]. Their main purpose is to reduce or eliminate the symptoms generated by myofascial trigger points (TrPs), which are defined as severely irritated areas within the hypertonic muscle fiber band or the fascia itself. Latent TrPs are described as those that do not generate symptoms on their own. However, they can cause refered pain at the time of provocation, i.e. pressure at the place of their occurrence.

In the scientific literature there are no reports on the assessment of the combination of MET with TPT

DETAILED DESCRIPTION:
The randomized study will focus on assessing the effectiveness of 3 different physiotherapeutic interventions. The physiotherapist with 10 years of professional experience will be responsible for performing all diagnostic procedures and therapeutic interventions.

Diagnosis of latent trigger point will be performed on subjects in the supine position. The therapist using a pincer grip will perform palpation in the area of the entire upper trapezius muscle. Testing for the presence of trigger point can be considered positive when it is noted: 1) the presence of a detectable strained band in the muscle, 2) the presence of an excessively sensitive area in the strained muscle band, 3) the response of local vibration caused by compression of the strained band, 4) occurrence of characteristic transferred symptoms (pain radiating to the posterior-lateral side of the neck, and/or mastoid process of the temporal bone, and/or the temporal bone area, and/or the angle of the jaw) as a result of compression of the hypersensitive muscle band. The test will be performed on both sides of this muscle.

The following measurement methods are planned to be used:

1. Electrogoniometry of the cervical spine. A Penny & Giles strain tensometric electrogoniometer will be used. Using this device, the angular values of cervical spine movements will be examined. The SG150 two-plane sensor and the Q110 single-plane sensor will be used. The lower edge of the upper sensor will be attached around the occipital tuberosity, while the upper edge of the lower sensor on the C7 spinous process. The examined person will be in a sitting position. Double-sided tape from Biometrics will be used to stick the electrogoniometer sensors. For the measurements of each movement, the subject will perform 3 repetitions. Then the mean value will be calculated, which will be the result.
2. Myotonometry. In order to examine the biophysical parameters of soft tissues a MyotonPRO will be used.

   Measurements will be made on the upper part of the trapezius muscle at the point located in the middle of the segment between the C7 spinous process and the shoulder angle of the acromion. During measurements, the subject will be lying down.
3. Pressure pain threshold (PPT). The Wagner Instruments Algometer will be used to assess the subjective parameter - pressure pain threshold of first discomfort. The place of measurement will be the point located on the upper trapezius muscle in the middle of the segment between the C7 spinous process and the shoulder angle of the acromion. The subject will be lying down on his back. Pressure from the algometer sensor will be applied from above and perpendicular to the examined muscle. Three measurements will be taken alternately for both sides of the upper trapezius. The mean value will be calculated, which will be the results for the right and left sides of the examined muscle.

The order of measurements will be: 1) myotometry, 2) pressure pain threshold test, 3) cervical spine electrogoniometry.

Participation in the study will be voluntary, free and fully anonymous. The participant will be able to opt out of the study at any stage. All planned therapeutic and measurement methods are non-invasive and safe. They do not threaten the health and life of the respondents.

ELIGIBILITY:
Inclusion Criteria:

* right-handed people
* amateur practicing symmetrical sports (eg. swimming, running, cycling, gym, roller skates)
* asymptomatic subjects (without pain symptoms of the cervical spine and shoulder girdle)
* occurrence of latent trigger point of the upper trapezius muscle

Exclusion Criteria:

* age above 21 years
* no latent trigger point on the upper trapezius muscle
* pain in the cervical spine or shoulder girdle
* any neurological symptoms in the upper limb
* previous operations in the cervical spine or shoulder girdle
* practicing asymmetrical sports
* professional sports

Ages: 19 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Cervical Anterior Flexion before the intervention | PRE (immediately before the intervention)
  Electrogoniometric measurement of the angular range of motion immediately before the intervention.
Cervical Anterior Flexion after the intervention | POST (immediately after the intervention)
  Electrogoniometric measurement of the angular range of motion immediately after the intervention.
Cervical Anterior Flexion on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Electrogoniometric measurement of the angular range of motion on the next day after the intervention.
Cervical Posterior Flexion before the intervention | PRE (immediately before the intervention)
  Electrogoniometric measurement of the angular range of motion immediately before the intervention.
Cervical Posterior Flexion after the intervention | POST (immediately after the intervention)
  Electrogoniometric measurement of the angular range of motion immediately after the intervention.
Cervical Posterior Flexion on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Electrogoniometric measurement of the angular range of motion on the next day after the intervention.
Cervical Right Flexion before the intervention | PRE (immediately before the intervention)
  Electrogoniometric measurement of the angular range of motion immediately before the intervention.
Cervical Right Flexion after the intervention | POST (immediately after the intervention)
  Electrogoniometric measurement of the angular range of motion immediately after the intervention.
Cervical Right Flexion on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Electrogoniometric measurement of the angular range of motion on the next day after the intervention.
Cervical Left Flexion before the intervention | PRE (immediately before the intervention)
  Electrogoniometric measurement of the angular range of motion immediately before the intervention.
Cervical Left Flexion after the intervention | POST (immediately after the intervention)
  Electrogoniometric measurement of the angular range of motion immediately after the intervention.
Cervical Left Flexion on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Electrogoniometric measurement of the angular range of motion on the next day after the intervention.
Cervical Right Rotation before the intervention | PRE (immediately before the intervention)
  Electrogoniometric measurement of the angular range of motion immediately before the intervention.
Cervical Right Rotation after the intervention | POST (immediately after the intervention)
  Electrogoniometric measurement of the angular range of motion immediately after the intervention.
Cervical Right Rotation on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Electrogoniometric measurement of the angular range of motion on the next day after the intervention.
Cervical Left Rotation before the intervention | PRE (immediately before the intervention)
  Electrogoniometric measurement of the angular range of motion immediately before the intervention.
Cervical Left Rotation after the intervention | POST (immediately after the intervention)
  Electrogoniometric measurement of the angular range of motion immediately after the intervention.
Cervical Left Rotation on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Electrogoniometric measurement of the angular range of motion on the next day after the intervention.
Stiffness (S) of the upper right trapezius muscle before the intervention | PRE (immediately before the intervention)
  Myotonometric examination of soft tissue properties immediately before the intervention.
Stiffness (S) of the upper right trapezius muscle after the intervention | POST (immediately after the intervention)
  Myotonometric examination of soft tissue properties immediately after the intervention.
Stiffness (S) of the upper right trapezius muscle on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Myotonometric examination of soft tissue properties on the next day after the intervention.
Stiffness (S) of the upper left trapezius muscle before the intervention | PRE (immediately before the intervention)
  Myotonometric examination of soft tissue properties immediately before the intervention.
Stiffness (S) of the upper left trapezius muscle after the intervention | POST (immediately after the intervention)
  Myotonometric examination of soft tissue properties immediately after the intervention.
Stiffness (S) of the upper left trapezius muscle on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Myotonometric examination of soft tissue properties on the next day after the intervention.
Elasticity (D) of the upper right trapezius muscle muscle before the intervention | PRE (immediately before the intervention)
  Myotonometric examination of soft tissue properties immediately before the intervention.
Elasticity (D) of the upper right trapezius muscle after the intervention | POST (immediately after the intervention)
  Myotonometric examination of soft tissue properties immediately after the intervention.
Elasticity (D) of the upper right trapezius muscle on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Myotonometric examination of soft tissue properties on the next day after the intervention.
Elasticity (D) of the upper left trapezius muscle before the intervention | PRE (immediately before the intervention)
  Myotonometric examination of soft tissue properties immediately before the intervention.
Elasticity (D) of the upper left trapezius muscle after the intervention | POST (immediately after the intervention)
  Myotonometric examination of soft tissue properties immediately after the intervention.
Elasticity (D) of the upper left trapezius muscle on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Myotonometric examination of soft tissue properties on the next day after the intervention.
Muscle tone (F) of the upper right trapezius muscle before the intervention | PRE (immediately before the intervention)
  Myotonometric examination of soft tissue properties immediately before the intervention.
Muscle tone (F) of the upper right trapezius muscle after the intervention | POST (immediately after the intervention)
  Myotonometric examination of soft tissue properties immediately after the intervention.
Muscle tone (F) of the upper right trapezius muscle on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Myotonometric examination of soft tissue properties on the next day after the intervention.
Muscle tone (F) of the upper left trapezius muscle before the intervention | PRE (immediately before the intervention)
  Myotonometric examination of soft tissue properties immediately before the intervention.
Muscle tone (F) of the upper left trapezius muscle after the intervention | POST (immediately after the intervention)
  Myotonometric examination of soft tissue properties immediately after the intervention.
Muscle tone (F) of the upper left trapezius muscle on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Myotonometric examination of soft tissue properties on the next day after the intervention.
Pressure pain threshold (PPT) of the upper right trapezius muscle before the intervention | PRE (immediately before the intervention)
  Examination of the first discomfort threshold using an algometer immediately before the intervention.
Pressure pain threshold (PPT) of the upper right trapezius muscle after the intervention | POST (immediately after the intervention)
  Examination of the first discomfort threshold using an algometer immediately after the intervention.
Pressure pain threshold (PPT) of the upper right trapezius muscle on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Examination of the first discomfort threshold using an algometer on the next day after the intervention.
Pressure pain threshold (PPT) of the upper left trapezius muscle before the intervention | PRE (immediately before the intervention)
  Examination of the first discomfort threshold using an algometer immediately before the intervention.
Pressure pain threshold (PPT) of the upper left trapezius muscle after the intervention | POST (immediately after the intervention)
  Examination of the first discomfort threshold using an algometer immediately after the intervention.
Pressure pain threshold (PPT) of the upper left trapezius muscle on the next day after the intervention | FOLLOW-UP (the next day after the intervention)
  Examination of the first discomfort threshold using an algometer on the next day after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Michał Wendt, PhD, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Department of Biology and Anatomy, Department of Motor Organ Rehabilitation, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
University IPD sharing platform is under preparation. All data will also be available to researchers via the principal researcher's email (wendt@awf.poznan.pl) or Research Gate website.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from June 2020.
Access Criteria: Available to all researchers
URL: http://www.awf.poznan.pl/pl/noz-anatomia-biologia-aktualnosci

REFERENCES:
- [Background] Ko CY, Choi HJ, Ryu J, Kim G. Between-day reliability of MyotonPRO for the non-invasive measurement of muscle material properties in the lower extremities of patients with a chronic spinal cord injury. J Biomech. 2018 May 17;73:60-65. doi: 10.1016/j.jbiomech.2018.03.026. Epub 2018 Mar 17. PMID 29599041
- [Background] Dellalana LE, Chen F, Vain A, Gandelman JS, Poldemaa M, Chen H, Tkaczyk ER. Reproducibility of the durometer and myoton devices for skin stiffness measurement in healthy subjects. Skin Res Technol. 2019 May;25(3):289-293. doi: 10.1111/srt.12646. Epub 2018 Nov 10. PMID 30414198
- [Background] Dissanayaka TD, Farrell M, Zoghi M, Egan GF, Jaberzadeh S. Test-retest reliability of subjective supra-threshold scaling of multiple pressure-pain sensations among healthy individuals: a study using hydraulic pressure algometry. Somatosens Mot Res. 2018 Sep-Dec;35(3-4):153-161. doi: 10.1080/08990220.2018.1505608. Epub 2018 Oct 9. PMID 30299201
- [Background] Chen Q, Wang HJ, Gay RE, Thompson JM, Manduca A, An KN, Ehman RE, Basford JR. Quantification of Myofascial Taut Bands. Arch Phys Med Rehabil. 2016 Jan;97(1):67-73. doi: 10.1016/j.apmr.2015.09.019. Epub 2015 Oct 14. PMID 26461163
- [Background] Vernon H, Schneider M. Chiropractic management of myofascial trigger points and myofascial pain syndrome: a systematic review of the literature. J Manipulative Physiol Ther. 2009 Jan;32(1):14-24. doi: 10.1016/j.jmpt.2008.06.012. PMID 19121461
- [Background] Clark BC, Thomas JS, Walkowski SA, Howell JN. The biology of manual therapies. J Am Osteopath Assoc. 2012 Sep;112(9):617-29. PMID 22984235
- [Background] Ribeiro DC, Belgrave A, Naden A, Fang H, Matthews P, Parshottam S. The prevalence of myofascial trigger points in neck and shoulder-related disorders: a systematic review of the literature. BMC Musculoskelet Disord. 2018 Jul 25;19(1):252. doi: 10.1186/s12891-018-2157-9. PMID 30045708
- [Background] Fernandez-de-las-Penas C, Dommerholt J. Myofascial trigger points: peripheral or central phenomenon? Curr Rheumatol Rep. 2014 Jan;16(1):395. doi: 10.1007/s11926-013-0395-2. PMID 24264721
- [Background] Giamberardino MA, Affaitati G, Fabrizio A, Costantini R. Myofascial pain syndromes and their evaluation. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):185-98. doi: 10.1016/j.berh.2011.01.002. PMID 22094195
- [Background] Ge HY, Fernandez-de-Las-Penas C, Yue SW. Myofascial trigger points: spontaneous electrical activity and its consequences for pain induction and propagation. Chin Med. 2011 Mar 25;6:13. doi: 10.1186/1749-8546-6-13. PMID 21439050
- [Result] Munoz-Munoz S, Munoz-Garcia MT, Alburquerque-Sendin F, Arroyo-Morales M, Fernandez-de-las-Penas C. Myofascial trigger points, pain, disability, and sleep quality in individuals with mechanical neck pain. J Manipulative Physiol Ther. 2012 Oct;35(8):608-13. doi: 10.1016/j.jmpt.2012.09.003. PMID 23158466
- [Result] Cagnie B, Dewitte V, Coppieters I, Van Oosterwijck J, Cools A, Danneels L. Effect of ischemic compression on trigger points in the neck and shoulder muscles in office workers: a cohort study. J Manipulative Physiol Ther. 2013 Oct;36(8):482-9. doi: 10.1016/j.jmpt.2013.07.001. Epub 2013 Aug 28. PMID 23993756
- [Result] Yoo WG. Comparison of the Symmetry of Right and Left Lateral Cervical Flexion and Rotation and the Cervical FRR in Young Computer Workers. J Phys Ther Sci. 2014 May;26(5):783-4. doi: 10.1589/jpts.26.783. Epub 2014 May 29. PMID 24926152
- [Result] Yeganeh Lari A, Okhovatian F, Naimi Ss, Baghban AA. The effect of the combination of dry needling and MET on latent trigger point upper trapezius in females. Man Ther. 2016 Feb;21:204-9. doi: 10.1016/j.math.2015.08.004. Epub 2015 Aug 14. PMID 26304789
- [Result] Sadria G, Hosseini M, Rezasoltani A, Akbarzadeh Bagheban A, Davari A, Seifolahi A. A comparison of the effect of the active release and muscle energy techniques on the latent trigger points of the upper trapezius. J Bodyw Mov Ther. 2017 Oct;21(4):920-925. doi: 10.1016/j.jbmt.2016.10.005. Epub 2016 Oct 21. PMID 29037649
- [Result] Kisilewicz A, Janusiak M, Szafraniec R, Smoter M, Ciszek B, Madeleine P, Fernandez-de-Las-Penas C, Kawczynski A. Changes in Muscle Stiffness of the Trapezius Muscle After Application of Ischemic Compression into Myofascial Trigger Points in Professional Basketball Players. J Hum Kinet. 2018 Oct 15;64:35-45. doi: 10.2478/hukin-2018-0043. eCollection 2018 Sep. PMID 30429897
- [Result] Mohammadi Kojidi M, Okhovatian F, Rahimi A, Baghban AA, Azimi H. The influence of Positional Release Therapy on the myofascial trigger points of the upper trapezius muscle in computer users. J Bodyw Mov Ther. 2016 Oct;20(4):767-773. doi: 10.1016/j.jbmt.2016.04.006. Epub 2016 Apr 7. PMID 27814857
- [Result] Bron C, Wensing M, Franssen JL, Oostendorp RA. Treatment of myofascial trigger points in common shoulder disorders by physical therapy: a randomized controlled trial [ISRCTN75722066]. BMC Musculoskelet Disord. 2007 Nov 5;8:107. doi: 10.1186/1471-2474-8-107. PMID 17983467
- [Result] Gross A, Kay TM, Paquin JP, Blanchette S, Lalonde P, Christie T, Dupont G, Graham N, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Hoving JL, Bronfort G, Santaguida PL; Cervical Overview Group. Exercises for mechanical neck disorders. Cochrane Database Syst Rev. 2015 Jan 28;1(1):CD004250. doi: 10.1002/14651858.CD004250.pub5. PMID 25629215
- [Result] Burns DK, Wells MR. Gross range of motion in the cervical spine: the effects of osteopathic muscle energy technique in asymptomatic subjects. J Am Osteopath Assoc. 2006 Mar;106(3):137-42. PMID 16585381